CLINICAL TRIAL: NCT00116155
Title: A Phase I/II Dose Finding Trial of the Intravenous Injection of CV787, a Prostate-Specific Antigen Cytolytic Adenovirus, in Patients With Hormone Refractory Metastatic Prostate Cancer
Brief Title: Trial of IV Injection of CV787 in Hormone Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV787-9902
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2005-06-28 (Estimated); Status verified 2005-06

CONDITIONS: Prostate Cancer
Keywords: Hormone Refractory Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: CV787 (CG7870)

SUMMARY:
This is a multi-center, open-label, dose finding study of CV787 adenovirus in patients with hormone refractory metastatic prostate cancer. Patients will receive treatment intravenously at one of up to nine dose levels, each containing three to six patients.

Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
To determine the safety, tolerability, and the maximum tolerated dose of CG7870 when administered intravenously to patients with progressive metastatic hormone refractory prostate cancer

SECONDARY OUTCOMES:
To evaluate prostate-specific antigen (PSA) response rates, duration of response, and time to disease progression
To evaluate other clinical efficacy responses observed
To evaluate the systemic pharmacokinetics of CG7870 after intravenous administration
To monitor the immune response to CG7870